CLINICAL TRIAL: NCT05512884
Title: Testing the Effect of Speeded Anomia Therapy in Patients With Chronic Post-stroke Aphasia: a Cross-over Randomized Controlled Trial
Brief Title: Speeded Anomia Treatment in Chronic Post-stroke Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Matthew A. Lambon Ralph, Professor, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 01/8/094
Record Dates: First submitted 2022-08-17; First posted 2022-08-23 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Aphasia
Keywords: Anomia; Speech Disorders; Language Disorders; Communication Disorders
MeSH Terms: conditions — Aphasia; Anomia; Speech Disorders; Language Disorders; Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speeded anomia therapy (Experimental): 21h of anomia therapy
  Interventions: Behavioral: Speeded anomia therapy
- Standard care (No Intervention): Participants' typical daily routine

INTERVENTIONS:
Behavioral: Speeded anomia therapy — The speeded anomia therapy was introduced as RISP (Repeated, Increasingly Speeded Production) by Conroy et al. (2018). Participants are asked to name the picture presented to them before an auditory stimulus ('beep' sound) at the end of item presentation. In each session the allotted response time is gradually reduced. After an incorrect response, participants are asked to repeat the word three times.
  Arms: Speeded anomia therapy

SUMMARY:
The main aim of the study is to investigate the effect of a novel, speeded anomia therapy (Conroy et al., 2018) in a large population of patients with chronic post-stroke aphasia. The treatment will be delivered via a web application (QuickWord).

DETAILED DESCRIPTION:
The main aim is to test the clinical efficacy of a novel, web based, rehabilitation approach to aphasic word-finding difficulties (QuickWord). In an initial development and case-series evaluation, Conroy et al (2018, Brain) found that training for both speed as well as accuracy of naming generated much better outcomes to picture naming accuracy and also augmented the carry-over to connected speech production.

This is a randomised, crossover, clinical trial of QuickWord in a group of aphasic patients in the chronic post-stroke period. The comparison will be standard care. The main outcome measures are clinically relevant improvement in naming to confrontation, and spontaneous use of the target vocabulary in a connected speech sample (detailed picture description). Secondary outcome includes measured use of the vocabulary in a story-telling, connected speech assessment (retelling of the Cinderella story).

ELIGIBILITY:
Inclusion Criteria:

* Native English speakers
* Age 18 years or above
* Stroke (any type) greater than 12 months post onset
* No history of neurological disorders / psychiatric disorders
* Normal or corrected-to-normal hearing & vision
* Able to give informed consent
* Currently not receiving Speech & Language therapy
* Minimal repetition skills (>40% on an immediate word repetition test)
* Evidence of naming difficulties (<90% in Boston Naming Test - Goodglass et al., 1983)

Exclusion Criteria:

* Non-native English speakers
* Less than 18 years old
* Stroke less than 12 months post onset
* History of neurological disorders / psychiatric disorders
* Uncorrected hearing & vision
* Unable to give informed consent
* Currently receiving Speech & Language therapy
* Insufficient repetition skills (<40% on an immediate word repetition test)
* Good naming performance (>90% in Boston Naming Test - Goodglass et al., 1983)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-15 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Speeded anomia therapy effect in reaction time | Measured over 10 weeks (Week 0, Week 2, Week 4, Week 6, Week 10)
  Change in reaction time in single-item picture naming
Speeded anomia therapy effect in accuracy | Measured over 10 weeks (Week 0, Week 2, Week 4, Week 6, Week 10)
  Change in accuracy in single-item picture naming
Generalisation to connected speech | Measured over 10 weeks (Week 0, Week 2, Week 4, Week 6, Week 10)
  Change in word retrieval in composite picture description. Participants will be asked to describe composite pictures (from the "Where's Waldo/Wally?" publications).

SECONDARY OUTCOMES:
Generalisation to story-telling connected speech | Measured over 10 weeks (Week 0, Week 2, Week 4, Week 6, Week 10)
  Change in narrative speech production. Participants will be asked to narrate the Cinderella story. A checklist with some of the most frequently used nouns (data obtained from AphasiaBank database) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lambon Ralph, DPhil, Principal Investigator — MRC Cognition and Brain Sciences Unit, University of Cambridge
Locations (1):
- MRC Cognition & Brain Sciences Unit, Cambridge, United Kingdom

REFERENCES:
- [Background] Conroy P, Sotiropoulou Drosopoulou C, Humphreys GF, Halai AD, Lambon Ralph MA. Time for a quick word? The striking benefits of training speed and accuracy of word retrieval in post-stroke aphasia. Brain. 2018 Jun 1;141(6):1815-1827. doi: 10.1093/brain/awy087. PMID 29672757